CLINICAL TRIAL: NCT05466201
Title: A Multicenter Clinical Study of a TPO Receptor Agonist (Eltrombopag) in the Acceleration of Engraftment Post Hematopoietic Stem Cell Transplantation of Bone Marrow Failure Diseases
Brief Title: The Use of Eltrombopag Post HSCT in BMFD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, HAN Yue, Principal Investigator, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SOOCHOW-HY-2022-08
Record Dates: First submitted 2022-07-12; First posted 2022-07-20 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Stem Cell Transplant Complications
Keywords: Hematopoietic stem cell transplantation; Bone marrow failure syndrome; Eltrombopag; Thrombocytopenia
MeSH Terms: conditions — Bone Marrow Failure Disorders; Thrombocytopenia | interventions — eltrombopag; Tablets; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- supportive care (Other): patients in this group will receive supportive care, including blood products transfusion, anti-infective therapy rather than rhTPO or TPO-RAs.
  Interventions: Drug: Supportive care
- Eltrombopag group (Experimental): Eltrombopag treatment will be started at the dose of 50mg/d from the 1st day post hematopoietic stem cell transplantation, and the dose will be titrated by 25mg each every 7 days up to 100mg/d according to the tolerability. If not tolerable, reduce the dose to the previous tolerable level (if not tolerable at 50mg/d, reduce to 25mg/d) and maintain this dose for the following 7 days, with the attempt to restart dose escalation after this 7-day period.
  Interventions: Drug: Eltrombopag 25 MG Oral Tablet

INTERVENTIONS:
Drug: Eltrombopag 25 MG Oral Tablet — Since thrombopoietin receptor agonists (TPO-RAs) have never been regularly used for promotion of cell engraftment post hematopoietic stem cell transplantation HSCT), we design this eltrombopag intervention to evaluate the safety and efficacy of TPO-RAs post HSCT.
  Other Names: TPO-RA
  Arms: Eltrombopag group
Drug: Supportive care — Patients receive transfusion of blood products, including platelets and red blood cells.
  Other Names: support
  Arms: supportive care

SUMMARY:
Bone marrow failure disease(BMFD) is a kind of bone marrow due to congenital or acquired hematopoietic stem cells (hemopoietic stem cell, HSC) function damage. Allogenic hemopoietic stem cell transplantation (Allo-HSCT) might be the most possible treatment to cure the disease.However, 5-26% of patients have been reported to have delayed platelet engraftment (DPE), which is defined as persistent severe thrombocytopenia (<20 × 109/L) for >35 days after transplantation . To date, no standard treatment and prevention has been recommended for DPE. In patients with DPE, the amount of transfusion, the increased risk of infection, and the prolonged average hospital stay were independent risk factors affecting the prognosis of allo-HSCT patients. Due to continuous and progressive failure in the bone marrow hematopoiesis, thrombocytopenia post HSCT is more common in BMFD patients and often achieves low response to conventional therapy, such as platelet transfusion. Therefore, it is of great significance to effectively promote hematopoietic reconstruction to improve the prognosis of transplant patients.

DETAILED DESCRIPTION:
Bone marrow failure disease(BMFD) is a kind of bone marrow due to congenital or acquired hematopoietic stem cells (hemopoietic stem cell, HSC) function damage. Generally, BMFD can be divided into two categories based on pathogenesis, which is primary and secondary BMFD. The latter is commonly seen secondary to infection, cancer, drugs, while aplastic anemia(AA), hypoplastic myelodysplastic syndromes(hMDS), paroxysmal nocturnal haemoglobinuria(PNH) and Fanconi anaemia(FA) are included in primary BMFD. Although immunotherapy or allogenic hemopoietic stem cell transplantation (Allo-HSCT) can be selected based on different individuals, allo-HSCT is still the most effective treatment for diseases that pose a greater threat to life or have a higher degree of malignancy, such as sereve aplastic anemia(SAA), MDS and PNH. Patients undergoing allo-HSCT typically achieve neutrophil and megakaryocyte reconstruction within 2 weeks and 3 weeks after transplantation respectively. However, 5-26% of patients have been reported to have delayed platelet engraftment (DPE), which is defined as persistent severe thrombocytopenia (<20 × 109/L) for >35 days after transplantation . To date, no standard treatment and prevention has been recommended for DPE. In patients with DPE, the amount of transfusion, the increased risk of infection, and the prolonged average hospital stay were independent risk factors affecting the prognosis of allo-HSCT patients. Due to continuous and progressive failure in the bone marrow hematopoiesis, thrombocytopenia post HSCT is more common in BMFD patients and often achieves low response to conventional therapy, such as platelet transfusion. Therefore, it is of great significance to effectively promote hematopoietic reconstruction to improve the prognosis of transplant patients.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed as bone marrow failure disease who received allo-HSCT; Physical strength score 0-3 according to WHO standard

Exclusion Criteria:

1. single or double umbilical cord blood transplantation;
2. allergic to any of the research drugs involved in the protocol;
3. simultaneously suffering from another malignant tumor;
4. pregnant or lactating women;
5. participating in other clinical researchers at the same time;
6. patients with at least one following high risk factors of thrombosis: past medical history of thromboembolism, concurrent grade 2 to 3 hypertension (systolic BP>=160mmHg or diastolic BP>=100mmHg) , diabetes, obesity(BMI>30), family history of stroke, smoke for more than 10 years , or history of catheter thrombosis;
7. severe cataract;
8. Severe infectious diseases (uncured tuberculosis, pulmonary aspergillosis, viral infection, active hepatitis B/C; for positive HBsAg and HBcAg, patient is excluded if hepatitis B DNA nucleic acid test is positive, DNA negative patients can enter this clinical trial; patients with hepatitis C who have a positive hepatitis C RNA nucleic acid test are excluded).;
9. Abnormal liver and kidney function: creatinine level ≥177 μmol/l (1.5mg/dl), transaminase and bilirubin levels increased significantly (3 times or more than the upper limit of normal), and who cannot be enrolled at the discretion of clinician.
10. In moribund condition or concurrent severe liver, kidney, heart, nerve, lung, infectious or metabolic diseases, the severity of which will cause the patient to be unable to tolerate the treatment regimen, or may die within 7-10 days

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2022-10-22 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Number and proportion of platelet engraftment on day 35 post HSCT. | From day 28 to 35 post HSCT
  Platelet engraftment is defined as platelet count >20×109/L in consecutive 7 days (namely day 28 to day 35 after HSCT) without platelet transfusion in the prior 7 days (in other words, no platelet transfusion after day 21).

SECONDARY OUTCOMES:
Number and proportion of subjects achieving neutrophil engraftment at day 35 post HSCT. | From day 28 to 35 post HSCT
  Neutrophil engraftment is defined as ANC>0.5×109/L for consecutive 3 days without administration of G-csf
Hematopoietic reconstruction time. | From day 1 to day 180 post HSCT
  Reconstruction time is defined as the time from day 1 after allo-HSCT to platelet or neutrophil engraftment
Overall survival (OS) | From day 1 to day 720 post HSCT or the time of the patients enrolled dead or quitting
  OS is defined as the time from the date of day 1 post HSCT to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, PhD,MD, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nash RA, Kurzrock R, DiPersio J, Vose J, Linker C, Maharaj D, Nademanee AP, Negrin R, Nimer S, Shulman H, Ashby M, Jones D, Appelbaum FR, Champlin R. A phase I trial of recombinant human thrombopoietin in patients with delayed platelet recovery after hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2000;6(1):25-34. doi: 10.1016/s1083-8791(00)70049-8. PMID 10707996
- [Background] Marotta S, Marano L, Ricci P, Cacace F, Frieri C, Simeone L, Trastulli F, Vitiello S, Cardano F, Pane F, Risitano AM. Eltrombopag for post-transplant cytopenias due to poor graft function. Bone Marrow Transplant. 2019 Aug;54(8):1346-1353. doi: 10.1038/s41409-019-0442-3. Epub 2019 Jan 24. PMID 30679824
- [Background] Mahat U, Rotz SJ, Hanna R. Use of Thrombopoietin Receptor Agonists in Prolonged Thrombocytopenia after Hematopoietic Stem Cell Transplantation. Biol Blood Marrow Transplant. 2020 Mar;26(3):e65-e73. doi: 10.1016/j.bbmt.2019.12.003. Epub 2019 Dec 9. PMID 31830528
- [Background] Zeidan AM, Battiwalla M, Berlyne D, Winkler T. Aplastic Anemia and MDS International Foundation (AAMDSIF): Bone marrow failure disease scientific symposium 2016. Leuk Res. 2017 Feb;53:8-12. doi: 10.1016/j.leukres.2016.11.011. Epub 2016 Nov 24. PMID 27923195
- [Background] Dominietto A, Raiola AM, van Lint MT, Lamparelli T, Gualandi F, Berisso G, Bregante S, Frassoni F, Casarino L, Verdiani S, Bacigalupo A. Factors influencing haematological recovery after allogeneic haemopoietic stem cell transplants: graft-versus-host disease, donor type, cytomegalovirus infections and cell dose. Br J Haematol. 2001 Jan;112(1):219-27. doi: 10.1046/j.1365-2141.2001.02468.x. PMID 11167808

DOCUMENTS (1):
  • Informed Consent Form (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT05466201/ICF_000.pdf